CLINICAL TRIAL: NCT03311243
Title: Effect of Non-surgical Periodontal Therapy on Systemic Inflammation in Thalassemia Major Patients With Chronic Periodontitis: A Randomised Controlled Clinical Trial
Brief Title: Periodontal Therapy in Thalassemia Major Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Saud University (Other)
Responsible Party: Principal Investigator, Zohaib Akram, Principal investigator, King Saud University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FR-17-67
Record Dates: First submitted 2017-10-11; First posted 2017-10-17 (Actual); Last update posted 2017-10-18 (Actual); Status verified 2017-10

CONDITIONS: Thalassemia Major; Chronic Periodontitis
Keywords: cytokines; scaling root planing; oral hygiene; systemic inflammation
MeSH Terms: conditions — beta-Thalassemia; Chronic Periodontitis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- β-Thalassemia major (TM- β) (Experimental)
  Interventions: Procedure: Non surgical periodontal therapy; Drug: Chemical plaque control
- Systemically healthy controls (Active Comparator)
  Interventions: Procedure: Non surgical periodontal therapy; Drug: Chemical plaque control

INTERVENTIONS:
Procedure: Non surgical periodontal therapy
Drug: Chemical plaque control

SUMMARY:
The study aims to evaluate the effect of local non surgical periodontal therapy on the systemic pro-inflammatory markers in the β-thalassemia (TM-β) patients with chronic periodontitis and systemically healthy demographically matched controls with chronic periodontitis. Both groups will receive non surgical periodontal therapy.

DETAILED DESCRIPTION:
Treatment modalities in patients with thalassemia include long-term transfusion therapy, iron chelation, splenectomy, allogeneic hematopoietic transplantation and supportive measures. Attempts to downgrade the systemic proinflammation and thereby reducing the morbidity of the disease warrants investigation in patients with β-thalassemia (TM-β). In blood disorders, as with most other diseases, achieving and maintaining inflammatory homeostasis is essential and necessary for survival. Both TM and gingival diseases cause increased levels of pro-inflammatory cytokines in the body fluids. Moreover, higher prevalence of gingival diseases is reported in children with TM. With oral hygiene maintenance and care, down-regulation of the systemic burden of the disease might be attained which will subsequently aid in achieving reduced morbidity in children with TM.

Both the groups will receive non surgical periodontal therapy (scaling and root planing) with the chlorhexidine containing adjunct in the form of a mouthrinse. Additionally, they will be taught standard tooth brushing technique (Fones technique). Participants will receive both verbal instructions and practical demonstrations.

ELIGIBILITY:
Inclusion Criteria:

1. Written and verbal consent
2. (TM-β) patients with gingivitis
3. Age: ≥10 years
4. Patients who have received or are receiving iron chelation therapy with deferasirox, calcium, vitamin D, and regular erythrocyte transfusion.

Exclusion Criteria:

1. Presence of hepatitis B or C or HIV-AIDS (Human immunodeficiency Virus- Acquired immunodeficiency syndrome).
2. Presence of any other known systemic disease.
3. Use of antibiotics or anti-inflammatory drugs within the past 6 months.
4. Dental prophylaxes in the last 6 months

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 52 (Actual)
Dates: Start 2016-01-11 (Actual); Primary Completion 2017-04-10 (Actual); Study Completion 2017-06-16 (Actual)

PRIMARY OUTCOMES:
Systemic pro-inflammatory cytokines | 6 weeks
  IL-6 and TNF-alpha potent proinflammatory cytokines

IPD SHARING:
Plan to Share IPD: Undecided